CLINICAL TRIAL: NCT05024929
Title: Targeted Therapy to Increase RAI Uptake in Patients With Metastatic Differentiated Thyroid Cancer
Brief Title: Targeted Therapy to Increase RAI Uptake in Metastatic DTC
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 21-018612
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Papillary Thyroid Cancer; Pediatric Cancer; Differentiated Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary; Neoplasms | interventions — Whole Body Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: Patients with differentiated thyroid cancer for whom oncogene-specific targeted therapy is planned from commercial supply or as part of a separate therapeutic trial
  Interventions: Procedure: Whole body scan
- Data Sharing Cohort: Patients with differentiated thyroid cancer enrolled on other oncogene-specific targeted therapy trials who undergo whole body thyroid scan approximately 28 days after beginning targeted therapy and agree to data sharing

INTERVENTIONS:
Procedure: Whole body scan — Patients will receive oncogene-specific molecularly targeted therapy independently of this protocol either via commercial supply of an FDA approved agent, or as part of a separate therapeutic clinical trial/compassionate use protocol/single patient investigational new drug (IND).
  During screening, patients will undergo a baseline RAI-whole body scan (WBS) to assess RAI-avidity of their tumor per standard of care. Following approximately 28 days of targeted therapy, the WBS will be repeated to determine whether this therapy is associated with an increase in RAI-avidity of their tumor.
  Groups: Prospective Cohort

SUMMARY:
Papillary thyroid cancer (PTC) is a common type of differentiated thyroid cancer (DTC) in children and represents the second most common cancer in adolescent females. Recently targeted drugs that block many of the genetic drivers of DTC have become available. While Investigators know that these drugs shrink DTC tumors in many cases, the impact on radioactive iodine (RAI) avidity has not been systematically studied.

DETAILED DESCRIPTION:
This is an observational cohort study that will enroll patients with DTC metastatic to the lungs who will receive oncogene-specific targeted therapy as part of routine clinical care or a separate therapeutic clinical trial. After approximately 4 weeks of therapy, patients will have a whole body scan to determine the change in RAI-avidity of their tumor from baseline. Subsequent therapy will be at the discretion of the treating physician or according to the therapeutic trial on which the patient is enrolled.

ELIGIBILITY:
Inclusion Criteria (Prospective Cohort):

1. Patients with a histologic diagnosis of differentiated thyroid cancer
2. Presence of an neurotrophic tyrosine kinase receptors (NTRK)-fusion, RET-fusion, anaplastic lymphoma kinase (ALK)-fusion, BRAF V600 mutation, BRAF-fusion or other targetable alteration identified in a Clinical Laboratory Improvement Amendments/College of American Pathologists (CLIA/CAP) laboratory
3. Anatomically evaluable disease on chest Computed tomography (CT) meeting oneo f the following criteria (obtained within 180 days of enrollment):

   1. multiple (10 or more) noncalcified solid pulmonary nodules visible on CT and/or
   2. enlarging, discrete pulmonary nodules visible on CT of any number consistent with metastatic disease
4. Patients for whom systemic therapy with an oncogene-specific kinase inhibitor is planned from commercial supply or as part of a separate therapeutic clinical trial (that does not include data sharing with this protocol)/compassionate access protocol/single patient investigational new drug (IND). Such agents include, but are not limited to:

   1. Larotrectinib, entrectinib, selitrectinib, and repotrectinib for NTRK fusions
   2. Selpercatinib and pralsetinib for RET fusions
   3. Crizotinib, lorlatinib, repotrectinib, and alectinib for ALK fusions
   4. Dabrafenib and/or trametinib for BRAF V600 mutations
   5. Oncogene-specific kinase inhibitors other than those specifically delineated above must be approved by the overall study PI prior to enrollment

Inclusion Criteria (Data Sharing Cohort):

1. Patients enrolled on other oncogene-specific targeted therapy trials who undergo whole body thyroid scan approximately 28 days after beginning targeted therapy and agree to data sharing as part of the consent process for that trial.

Exclusion Criteria (All Cohorts):

1. No prior oncogene-specific targeted therapy allowed. However, patients may enroll within 4 weeks of starting oncogene-specific therapy if a pre-therapy WBS is available. Prior therapy with non-oncogene specific multi-thyrosine kinase inhibitors (such as sorafenib, lenvatinib, and/or cabozantanib) is allowed.
2. Females who are pregnant or breastfeeding are excluded due to the potential risks of the RAI used in the WBS to the fetus/neonate.
3. Patients who require sedation/general anesthesia to complete a WBS are excluded.
4. U.S. Military Personnel are excluded due to the Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) requirements.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll children and adolescents with differentiated thyroid cancer with pulmonary metastases who are planned to receive oncogene-specific targeted therapy.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2021-07-16 (Actual); Primary Completion 2031-02-01 (Estimated); Study Completion 2033-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with increased tumor RAI-avidity after receiving oncogene-specific, targeted therapy | up to 5 years
  The primary outcome measure is to determine the proportion of patients with differentiated thyroid cancer metastatic to the lungs for whom oncogene-specific, targeted therapy increases tumor RAI-avidity.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Children's Hospital Westmead, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No